CLINICAL TRIAL: NCT05293600
Title: Treating Residual OSA With Endotype-directed Pharmacotherapy (Aim 3)
Brief Title: Rescue Pharmacotherapy for OSA
Acronym: RescOSA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Andrew Wellman, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022p000430
Record Dates: First submitted 2022-02-23; First posted 2022-03-24 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Acetazolamide; Trazodone; Atomoxetine Hydrochloride; Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): This is a two arm study. Patients will receive only one of the following drugs based on their altered sleep apnea trait. Patients with decreased arousal threshold will undergo treatment with placebo or Trazodone 100 mg in random order (one pill before 30 minutes before bedtime), patients with decreased pharyngeal muscle responsiveness will undergo treatment with placebo or Atomoxetine 80 mg + Eszopiclone 3 mg in random order (one pill before 30 minutes before bedtime), patients with increased loop gain will undergo treatment with placebo or Acetazolamide 500 mg in random order (one pill before 30 minutes before bedtime).
  Interventions: Drug: Placebo
- Interventional arm (Active Comparator): This is a two arm study. Patients will receive only one of the following drugs based on their altered sleep apnea trait. Patients with decreased arousal threshold will undergo treatment with placebo or Trazodone 100 mg in random order (one pill before 30 minutes before bedtime), patients with decreased pharyngeal muscle responsiveness will undergo treatment with placebo or Atomoxetine 80 mg + Eszopiclone 3 mg in random order (one pill before 30 minutes before bedtime), patients with increased loop gain will undergo treatment with placebo or Acetazolamide 500 mg in random order (one pill before 30 minutes before bedtime).
  Interventions: Drug: Acetazolamide; Drug: Trazodone; Drug: Atomoxetine and eszopiclone

INTERVENTIONS:
Drug: Placebo — Placebo capsule 30 min before bedtime
  Arms: Placebo
Drug: Acetazolamide — The intervention drug will be determined based on altered endotype and administered 30 min before bedtime. Patients will only take one drug of this intervention, which will be subsequently compared to placebo. Patients with increased loop gain will be given Acetazolamide 500 mg.
  Arms: Interventional arm
Drug: Trazodone — The intervention drug will be determined based on altered endotype and administered 30 min before bedtime. Patients will only take one drug of this intervention, which will be subsequently compared to placebo. Patients with decreased arousal threshold will be given Trazodone 100 mg.
  Arms: Interventional arm
Drug: Atomoxetine and eszopiclone — The intervention drug will be determined based on altered endotype and administered 30 min before bedtime. Patients will only take one drug of this intervention, which will be subsequently compared to placebo. Patients with decreased muscle responsiveness will be given Atomoxetine and Eszopiclone 80 + 3 mg.
  Arms: Interventional arm

SUMMARY:
Persistent obstructive sleep apnea (OSA) is common in people treated with mandibular advancement device (MAD) or hypoglossal nerve stimulation (HGNS). For most patients, these treatments are the last line of defense. If MAD or HGNS do not work, then patients are left to suffer the consequences of undertreated OSA. In this study, the investigators want to test the addition of a drug treatment to their regimen. Endotypes will be targeted pharmacologically with one of the following drugs: acetazolamide for a high loop gain, atomoxetine-plus-eszopiclone for poor pharyngeal muscle compensation, or trazodone for a low arousal threshold.

This aim is expected to provide treatment strategies for rescuing non-responders to MAD or HGNS therapy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have failed MAD or HGNS therapy, defined as a residual AHI ≥ 15 events/hr on MAD or HGNS therapy.

Exclusion Criteria:

* Sleep disordered breathing or respiratory disorders other than obstructive sleep apnea:

central sleep apnea (>50% of respiratory events scored as central), chronic hypoventilation/hypoxemia (awake SaO2 < 92% by oximetry) due to chronic obstructive pulmonary disease or other respiratory conditions.

* Other sleep disorders: periodic limb movements (periodic limb movement index > 20/hr), narcolepsy, or parasomnias.
* Any unstable major medical condition.
* Medications expected to stimulate or depress respiration (including opioids, barbiturates, benzodiazepines, doxapram, almitrine, theophylline, 4-hydroxybutanoic acid).
* Use of SSRIs/SNRIs.
* Contraindications for atomoxetine, including:
* pheochromocytoma
* use of monoamine oxidase inhibitors
* benign prostatic hypertrophy, urinary retention
* untreated narrow angle glaucoma
* bipolar disorder, mania, psychosis
* clinically significant constipation, gastric retention
* pre-existing seizure disorders
* clinically-significant kidney disorders
* clinically-significant liver disorders
* clinically-significant cardiovascular conditions
* severe hypertension (SBP>180 mmHg or DBP>110 mmHg measured at baseline)
* cardiomyopathy (LVEF<50%) or heart failure
* advanced atherosclerosi
* history of cerebrovascular events
* history of cardiac arrhythmias e.g., atrial fibrillation, QT prolongation
* other serious cardiac conditions that would raise the consequences of an increase in blood pressure or heart rate
* myasthenia gravis
* pregnancy/breast-feeding
* Contraindications for eszopiclone, including:
* Hypersensitivity to eszopiclone
* Chronic Obstructive Pulmonary Disease (COPD)
* Pregnancy
* Breast feeding
* Liver disease
* Contraindications for acetazolamide, including:
* Hyperchloremic acidosis
* Hypokalemia
* Hyponatremia
* Adrenal insufficiency
* Impaired kidney function
* Hypersensitivity to acetazolamide or other sulfonamides.
* Marked liver disease or impairment of liver function, including cirrhosis.
* Contraindications for trazodone, including:
* suicidal ideation
* bipolar disorder, mania
* use of monoamine oxidase inhibitors
* coronary artery disease
* cardiac arrhythmias
* QT prolongation
* hepatic disease
* renal failure or impairment
* closed angle glaucoma
* priapism
* pregnancy/breast-feeding

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI, Events/Hour of Sleep) | 1 night
  Based on previous studies the investigators anticipate that the interventional arm will reduce AHI through a positive effect on the abnormal endotype.

SECONDARY OUTCOMES:
Nadir oxygen saturation during sleep (LSpO2, %) | 1 night
  Based on previous studies the investigators anticipate that the interventional arm will reduce LSpO2 through a positive effect on the abnormal endotype.
Arousal Index (AI, Events/Hours of Sleep) | 1 night
  Based on previous studies the investigators anticipate that the interventional arm will reduce AI through inducing less fragmented sleep, which will be driven by a positive effect on the abnormal endotype.

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Disorders Research Program Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes